CLINICAL TRIAL: NCT01501825
Title: A Prospective, Comparative Study to Explore the Efficacy and Safety of the Five Channels Multiway Deep Transcranial Magnetic Stimulation (TMS) Device in Subjects With Major Depression Disorder (MDD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shalvata Mental Health Center (Other)
Collaborators: Brainsway-moach Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sha-16-11
Record Dates: First submitted 2011-12-27; First posted 2011-12-29 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2011-12

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- single channel (Active Comparator): Single Channel with a coil placed over the left PFC (10 Hz).
  Interventions: Device: 5 channels Multiway deep Transcranial Magnetic Stimulator
- four channels (Experimental): Four channels:
  1. 10 Hz over the left PFC.
  2. 1 Hz over the right PFC.
  3. 10 Hz over the left parietal cortex.
  4. 1 Hz over the right parietal cortex.
  Interventions: Device: five channels Multiway deep Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: 5 channels Multiway deep Transcranial Magnetic Stimulator — During the single channel treatment trial period the patients will receive the following dose of rTMS: 10 Hz - left DLPFC ( 10 Hz, at 120% MT, 3 sec pulse train, 20 second inter-train interval, 55 trains, i.e. a total of 1650 pulses per session, a total of 20 sessions in the study and a cumulative exposure (total number of pulses) of 33,000pulses in 4 weeks)
  Arms: single channel
Device: five channels Multiway deep Transcranial Magnetic Stimulation — During the four channels treatment trial period the patients will receive the following dose of rTMS: 10 Hz- left DLPFC, 1Hz - right DLPFC together, and than 10 Hz- left parietal cortex, 1Hz - right parietal cortex together.
  10 Hz protocol: ( 10 Hz, at 120% MT, 3 sec pulse train, 20 second inter-train interval, 55 trains, i.e. a total of 1650 pulses per session, a total of 20 sessions in the study and a cumulative exposure (total number of pulses) of 33,000pulses in 4 weeks)
  1 Hz protocol:
  1 Hz, at 120% MT, 5 min pulse train, 1 min inter-train interval, 6 trains, i.e. a total of 1800 pulses per session, a total of 20 sessions in the study and a cumulative exposure (total number of pulses) of 36,000 pulses in 4 weeks)
  Arms: four channels

SUMMARY:
The Multiway stimulator is a novel TMS stimulator with several new and unique properties. Currently standard TMS devices include a single channel, and can operate only a single coil. The Multiway stimulator includes five channels which can operate up to five independent TMS coils, either simultaneously or sequentially.

The Multiway device may be used to obtain a differential activation of various brain regions. For instance it can be used to induce high frequency stimulation of a certain brain region, thus inducing facilitation, while simultaneously stimulate at low frequency in another brain region, leading to inhibition.

The purpose of the study is to explore the efficacy and safety of Multiway deep TMS in comparison to a single channel DTMS treatment in subjects with MDD.

Subjects will be treated with one of two designs of the study device (the Multiway Coil TMS Device):

1. Single Channel with a coil placed over the left PFC (10 Hz).
2. Four channels: a. 10 Hz over the left PFC. b. 1 Hz over the right PFC. c. 10 Hz over the left parietal cortex. d. 1 Hz over the right parietal cortex.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient
* Diagnosed by senior psychiatrist as suffering from major depression episode according to DSM IV using the Structured Clinical Interview for DSM-4 (SCID).
* Rating on HDRS-21>20.
* Age: 18-68 years.
* Treated for the current depressive episode, at least four weeks, with at least one antidepressant in accepted dose, without improvement, according to their medical chart and ATHF ( antidepressant treatment history form) instruction guidelines .
* Gave informed consent for participation in the study.
* Negative answers on safety screening questionnaire for transcranial magnetic stimulation.

Exclusion Criteria:

* Diagnosis as suffering from other diagnosis on axis 1 ( like: schizophrenia, bipolar disorder, psychotic depression, geriatric depression).
* Diagnosis as suffering from Severe Borderline Personality Disorder or hospitalized due to exacerbation related to of borderline personality disorder.
* Substantial suicidal risk as judged by the treating psychiatrist.
* Attempted suicide in the past year.
* Any current unstable medical or surgical illness.
* History of seizure or heat convulsion.
* History of epilepsy or seizure in first degree relatives.
* History of head injury.
* History of any metal in the head (outside the mouth).
* Known history of any metallic particles in the eye, implanted cardiac pacemaker or any intracardiac lines, implanted neurostimulators, surgical clips, cochlear implants or any medical pumps.
* History of hearing loss.
* History of drug abuse or alcoholism in the last 6 month.
* Pregnancy or not using a reliable method of birth control.
* Systematic and metabolic unstable disorders.
* Inadequate communication with the patient.
* Under custodial care.
* Participation in current clinical study or clinical study within 30 days prior to this study.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Clinical antidepressant response | day 20
  Clinical antidepressant response at the end of the treatment, defined as a decline in Hamilton depression rating scale (HDRS-21) from the baseline rating by 50%.

SECONDARY OUTCOMES:
Clinical antidepressant remission | day 20
  Clinical antidepressant remission at the end of the treatment, define as exit HDRS-21 <10.
Symptomatic improvement | day 20
  Symptomatic improvement at the 4-week end point as measured with Hamilton Anxiety Rating Scale ( HARS), Quick Inventory of Depressive Symptomatology - Self Report (QIDS-SR) , Clinical Global Impression (CGI), Cognitive improvement measured by a computerized battery of tests (CANTAB).

CONTACTS AND LOCATIONS:
Overall Officials: Yechiel Levkovitz, MD, Phd, Principal Investigator — Shalvata Medical Health Center
Locations (2):
- Israel (2):
  - Shalvata Mental Health Center, Hod HaSharon
  - shalvata MHC, Hod HaSharon